CLINICAL TRIAL: NCT03863847
Title: A Neurofeedback Treatment for Chronic Musculoskeletal Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Natalie Mrachacz-Kersting, Associate Professor, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-20140041
Record Dates: First submitted 2019-01-02; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Chronic Musculoskeletal Pain; Tennis Elbow; Musculoskeletal Pain; Lateral Epicondylitis
Keywords: Pain; Chronic Pain; Musculoskeletal Pain; Treatment; Neurofeedback; Brain Activity; Brain Oscillation; Brain Computer Interface
MeSH Terms: conditions — Tennis Elbow; Musculoskeletal Pain; Pain; Chronic Pain | interventions — Neurofeedback; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Neurofeedback (Active Comparator): This intervention entails online feedback of pain-related neuronal oscillation power, and will be visualized to the individual for patient training purposes and for the eventual self-control of this brain activity.
  Interventions: Procedure: Neurofeedback
- Online Sham Neurofeedback (Sham Comparator): This intervention entails online sham feedback of non-pain related neuronal oscillation power, and will be visualized to the individual for patient training purposes and for the eventual self-control of this brain activity.
  Interventions: Procedure: Sham

INTERVENTIONS:
Procedure: Neurofeedback — The patients will receive neurofeedback on pain related brain-activity, and through training, learn to control said brain-activity.
  Arms: Online Neurofeedback
Procedure: Sham — The patients will receive sham neurofeedback on non-pain related brain-activity, and through training, learn to control said brain-activity.
  Arms: Online Sham Neurofeedback

SUMMARY:
This study evaluates the effects of a novel neurofeedback treatment on pain specific brainwaves in adults.

Chronic pain patients enrolled in this study will be randomized into a treatment group and a sham group.

DETAILED DESCRIPTION:
Recent research has underlined that central nervous system structures play a key role in the development of pain with significant maladaptive plasticity occurring in several brain areas. Non-pharmacological treatments, such as neurofeedback, are designed to restore normal brain function alongside with relieving pain symptoms. With a neurofeedback approach, the patient is provided with a feedback on specific brain waves recorded using non-invasive recording techniques (electroencephalography - EEG) and visualized on a screen.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from chronic pain due to tennis elbow for at least 3 months
* A clinical diagnosis of chronic lateral epicondylalgia,
* Pain associated with functional activities such as gripping and pain with resisted contraction of the wrist extensors or extensor carpi radialis brevis, or with passive stretching of the wrist extensors.

Exclusion Criteria:

* Clinical diagnosis of chronic lateral epicondylalgia on both sides, cervicothoracic spinal pathology, other upper limb musculoskeletal disorders or neurological disorders
* Pregnancy
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Previous or current neurologic, musculoskeletal or mental illnesses defined as an on-going systemic condition
* Lack of ability to cooperate
* Current use of medications that may affect the trial e.g. analgesics, anti- inflammatory drugs
* Consumption of alcohol, caffeine, nicotine or painkillers throughout the study period
* Past history of chronic pain, neurological or psychiatric conditions
* Participation in other pain trials throughout the study period and one month prior to participation
* Participation in more than two sessions of muscle training exercises per week involving the upper limb and/or lower back
* Evidence of other sources of elbow pain such as exacerbation of pain with neck movement or manual examination
* Sensory disturbances
* History of fractures
* Elbow surgery
* Contraindications to the use of TMS

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Up to three months
  Numerical pain scale ranging from 0 being no pain to 10 being worst imaginable pain (significant change in VAS score will be set to 1 at P = 0.05)

SECONDARY OUTCOMES:
Electroencephalographic (EEG) measurement. International 10-20 electrode placement with 10 channels placed on the contralateral hemisphere to the dominant limb being tested. | Up to three months
  Quantitative brain activity analysis to provide the subject with real-time feedback of their brain activity. The neurofeedback group will receive feedback on alpha brainwave power and learn to control this, while the sham group will receive feedback on non-pain related brain activity.
Electromyographic (EMG) measurement. | Up to three months
  EMG electrodes will be applied to the Extensor Carpi Radials Brevis (ECRB) muscle, to provide movement temporal features for EEG extraction.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Mrachacz Kersting, Dr, Study Director — Aalborg University, Department of Health Science and Technology
Locations (1):
- Center For Sensory-Motor Interaction, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No
Currently this study is under IP at Aalborg University and thus data cannot be shared at this point.